CLINICAL TRIAL: NCT04710186
Title: The Influence of Androgen Receptor, Insulin Like Growth Factor 1 Receptor, and Insulin Receptor in Male Patients With Peripheral Artery Disease
Brief Title: AR, IGF-IR, IR and Peripheral Artery Disease
Acronym: ANIMALPAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.39
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Androgen Receptor Abnormal; Insulin-Like Growth Factor I Deficiency; Insulin Receptor, Defect in
Keywords: peripheral artery disease; androgen receptor; Insulin-Like Growth Factor I; Insulin Receptor; Male
MeSH Terms: conditions — Insulin-Like Growth Factor I Deficiency; Insulin Receptor, Defect in; Peripheral Arterial Disease; Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male patients with PAD: The cohort was built to collect information about the role of androgen receptor, insulin receptor and Insulin-like Growth Factor 1 Receptor (IGF-IR) expression in patients with peripheral artery disease referred to Vascular Surgeon Specialist.
  Interventions: Procedure: arterial reconstructive open surgery

INTERVENTIONS:
Procedure: arterial reconstructive open surgery — Patients with peripheral artery disease (PAD) will undergo arterial reconstructive open surgery. Samples obtained from diseased arteries of lower limbs of patients undergoing arterial reconstructive open surgery will be collected and immediately preserved at -80°. Briefly, arterial tissues were excised, homogenized using a motor driven homogenizer and total RNA was isolated using Trizol reagent (Invitrogen, Milan, Italy), in accordance with the manufacturer's instructions. The expression of Androgen Receptor (AR), insulin receptor (IR) and the IGF-I receptor (IGF-IR) will be quantified by real-time PCR using platform Quant Studio7 Flex Real-Time PCR System (Thermo Fisher Scientific, Milan, Italy), following the manufacturer's instructions.

SUMMARY:
Peripheral artery Disease (PAD) is a major cardiovascular disease that can impair quality of life (QoL). It affects more often male patients and its pathophysiology is not completely known. Probably androgen receptors and metabolism alteration may play an important role in the onset and in the progression of PAD towards its dreadful complications. The aim of this study is to evaluate the role of Androgen Recetpr , IGF-I receptor, and Insulin Receptor on the arterial wall of male patients with PAD undergoing open revascularization surgery.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) of lower limbs is one of the most common clinical manifestation of atherosclerosis and can be considered a major cardiovascular disease with important morbidity and mortality, affecting also quality of life (QoL), thus representing an important public health concern. From a clinical point of view, PAD may be initially symptomatic with intermittent claudication (IC), and in critical limb ischemia (CLI), an advanced stage of PAD, with rest pain, and also with leg skin ulceration, a complication that may even lead to limb loss for amputation. From a pathophysiological point of view, in the presence of atherosclerosis, endothelial activation and dysfunction lead to hemodynamic alterations such as turbulent flow, abnormal shear stress, loss of potential energy, anomalies of vascular tone with functional impairment during leg exercise in early stages, with IC onset, and in advanced stages, during CLI stage, also with rest pain as a result of an important demand/perfusion mismatch. Endothelial dysfunction, and vascular tone are also regulated by sex hormones, and incidence and prevalence of PAD have usually been found to be higher in men than in women, and, more in general, males have a higher risk of developing cardiovascular disease during the reproductive period in comparison with females of the same age. This sex related difference in developing the disease was hypothesized to be related to the protective role of estrogens in female subjects, and harmful effects of androgens in male individuals. Furthermore, the androgen receptor (AR) seems to have a role in neointima formation, in influencing the size and the composition of atherosclerotic plaques, and also vascular smooth muscle cells (VSMCs) activity. Moreover, sex-specific effects on the metabolic system are well-known and associated with different risk profiles for cardiovascular disease and they have been also related to differences in sex hormones activities. In fact, the insulin and IGF-I signaling is mediated by hormone interaction with the insulin receptor (IR) and the IGF-I receptor (IGF-IR) which are members of subclass II of the tyrosine kinase receptor super-family and they, on one hand, participate to the metabolic homeostasis, and on the other hand, they have a direct role on VMMCs, and also in some stages of the atherosclerotic process..

The aim of this study is to evaluate the role of AR, IGF-IR, and IR on the arterial wall of male patients with PAD undergoing open revascularization surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with peripheral artery disease (PAD) eligible to receive arterial reconstructive open surgery.

Exclusion Criteria:

* active malignancy
* advanced liver disease
* advanced heart disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Inclusion criteria were patients with age >18 years, severe peripheral artery disease that needs surgical repair. Patients with life expectancy <6 months, advanced liver or heart disease and active malignancies were excluded. At the moment of hospital admission, clinicians collected the medical history including previous cardiovascular disease (CVD: stroke, coronary heart disease, heart failure, peripheral vascular disease), presence of dysmetabolism, history of arterial hypertension and diabetes, previous amputation, history of chronic kidney disease (CKD). Therapies practiced at home, encompassing hypoglycemic oral agents, insulin, blood pressure lowering drugs, statins, antiplatelet and anticoagulants were also collected.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Expression of AR, IGF-IR, IR | at 1year
  The expression of IR, IGF-IR and AR was quantified by real-time PCR using platform Quant Studio7 Flex Real-Time PCR System (Thermo Fisher Scientific, Milan, Italy), following the manufacturer's instructions

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Principal Investigator — University Magna Graecia of Catanzaro; Marcello Maggiolini, M.D., Study Chair — UNICAL - University of Calabria
Locations (1):
- University Magna Graecia of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song P, Rudan D, Zhu Y, Fowkes FJI, Rahimi K, Fowkes FGR, Rudan I. Global, regional, and national prevalence and risk factors for peripheral artery disease in 2015: an updated systematic review and analysis. Lancet Glob Health. 2019 Aug;7(8):e1020-e1030. doi: 10.1016/S2214-109X(19)30255-4. PMID 31303293
- [Background] Ielapi N, Licastro N, Catana M, Bracale UM, Serra R. Vascular Nursing and Vascular Surgery. Ann Vasc Surg. 2020 Oct;68:522-526. doi: 10.1016/j.avsg.2020.05.038. Epub 2020 May 29. PMID 32479881
- [Background] Orshal JM, Khalil RA. Gender, sex hormones, and vascular tone. Am J Physiol Regul Integr Comp Physiol. 2004 Feb;286(2):R233-49. doi: 10.1152/ajpregu.00338.2003. PMID 14707008
- [Background] Chistiakov DA, Myasoedova VA, Melnichenko AA, Grechko AV, Orekhov AN. Role of androgens in cardiovascular pathology. Vasc Health Risk Manag. 2018 Oct 15;14:283-290. doi: 10.2147/VHRM.S173259. eCollection 2018. PMID 30410343
- [Background] Baars A, Oosting A, Lohuis M, Koehorst M, El Aidy S, Hugenholtz F, Smidt H, Mischke M, Boekschoten MV, Verkade HJ, Garssen J, van der Beek EM, Knol J, de Vos P, van Bergenhenegouwen J, Fransen F. Sex differences in lipid metabolism are affected by presence of the gut microbiota. Sci Rep. 2018 Sep 7;8(1):13426. doi: 10.1038/s41598-018-31695-w. PMID 30194317
- [Background] Beneit N, Fernandez-Garcia CE, Martin-Ventura JL, Perdomo L, Escribano O, Michel JB, Garcia-Gomez G, Fernandez S, Diaz-Castroverde S, Egido J, Gomez-Hernandez A, Benito M. Expression of insulin receptor (IR) A and B isoforms, IGF-IR, and IR/IGF-IR hybrid receptors in vascular smooth muscle cells and their role in cell migration in atherosclerosis. Cardiovasc Diabetol. 2016 Dec 1;15(1):161. doi: 10.1186/s12933-016-0477-3. PMID 27905925